CLINICAL TRIAL: NCT02535975
Title: The Effects of Metformin in Patients With Mild Graves' Ophthalmopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2014-0706
Record Dates: First submitted 2015-08-12; First posted 2015-08-31 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Mild Graves' Ophthalmopathy
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental): Metformin 500mg PO three times a day for 24 weeks
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo tab. PO three times a day for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Tablets metformin 500 mg PO three times a day for 24 weeks
  Arms: Metformin
Drug: Placebo — Tablets placebo PO three times a day for 24 weeks
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, double-blind, placebo-controlled study about the effect of metformin in patients with mild Graves' ophthalmopathy. Eighty patients with mild ophthalmopathy will be included. Each patient will be given either metformin (500mg PO three times a day) or placebo ( PO three times a day ) for 6 months and then followed for 6 months after withdrawal of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years
2. Patients should not have diabetes (HbA1c level at screening should be lower than 6.5)
3. Mild Graves' ophthalmopathy according to EUGOGO statement.
4. Clinical activity score lower than 4
5. Being euthyroid for at least 2 month before the enrollment
6. No previous specific therapy for GO in 6 month before the enrollment except for local measures (e.g. eye drops)

Exclusion Criteria:

1. Moderate-severe Graves' ophthalmopathy
2. Clinical activity score ≥ 4
3. Contraindication for metformin use as following: renal dysfunction (creatinine level should be within normal range), liver dysfunction (AST and ALT levels should be within normal range), severe concomitant illness
4. Pregnant women
5. Current use of metformin or containing preparations
6. Metformin intolerance
7. Inability to comply with the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-12; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Change of Clinical Activity Score (CAS) score | At 0, 6 and 12 months
  Comparison of CAS scores before and after treatment in each arm and an inter-arm
Change of NOSPECS score | At 0, 6 and 12 months
  Comparison of NOSPECS scores before and after treatment in each arm and an inter-arm.

SECONDARY OUTCOMES:
adverse events | At 0, 6 and 12 months
  Comparison of adverse events rate in each arm and an inter-arm.
Quality of life questionnaires (GO-QoL) | At 0, 6 and 12 months
  Comparison of Graves' ophthalmopathy Quality of life questionnaire (GO-QOL) scores before and after treatment in each arm and an inter-arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrinology, Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea